CLINICAL TRIAL: NCT03385317
Title: Mindfulness to Mitigate the Effect of Anxiety-depression-fear in COPD
Brief Title: Mindfulness to Mitigate the Effect of Anxiety-depression-fear in Chronic Obstructive Pulmonary Disease (COPD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There was not enough manpower to complete the study.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Roberto P. Benzo, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-007994
Record Dates: First submitted 2016-03-17; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness (Experimental)
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness

SUMMARY:
People with COPD have a greater risk for symptoms of depression, anxiety, and fear of breathlessness. Those emotions are independently associated with lower physical activity, poorer quality of life, and higher hospitalization and exacerbations; all independent predictors of survival and costs. There is a lack of treatment options to be routinely used in primary clinics for patients with COPD. Systematic reviews suggest that interventions that promote an accepting mode of response, such as mindfulness, might be more appropriate and effective for managing psychological distress in COPD patients, especially breathing-related anxiety.

Hypothesis: A home-based 8-week Mindfulness-Based Stress Reduction (MBSR) for COPD targeted to individuals with symptoms of depression, anxiety, or fear of breathlessness delivered by a mindfulness coach using a combination of in-person sessions and remote video call sessions will be effective in improving emotional and overall quality of life, and measured physical activity.

ELIGIBILITY:
Inclusion criteria:

* Lung disease diagnosis
* Demonstrated competence in proposed technology
* Current or past smoking status
* Patient Health Questionnaire-2 (PHQ-2) or Generalized Anxiety Disorder scale (GAD-2) score >2 points or answering yes to a validated question of fear of being breathless ("Do you experience fear, or panic when you have difficulty getting your breath a good bit of the time?")

Exclusion criteria:

* High likelihood of non-compliance or low confidence using the technology
* Patients currently in pulmonary rehabilitation
* Inability to walk
* Prescribed antidepressant or antianxiety medication within last month
* Documented substance abuse
* Cognitive impairment as defined by the Mini-Mental test score < 24.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life as measured by the Chronic Respiratory Questionnaire | baseline, 20 weeks
  The Chronic Respiratory Disease Questionnaire is a disease-specific health-related quality of life questionnaire. It was developed to measure the impact of Chronic Obstructive Pulmonary Disease (COPD) on a person's life. It consists of 20 items across four dimensions: dyspnea, fatigue, emotional function, and mastery. Items in each section are scored from 1 (most severe) to 7 (no impairment). Therefore total scores can range from 20 (severe impairment) to 140 (no impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Benzo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No